CLINICAL TRIAL: NCT02643121
Title: Diagnostic and Prognostic Utility of Presepsin for Sepsis and Systemic Inflammatory Response Syndrome in Children
Brief Title: Utility of Presepsin in Children Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Jiří Žurek, M.D., Ph.D., Brno University Hospital
Other Study IDs: KDAR 19 - 1
Record Dates: First submitted 2015-12-08; First posted 2015-12-31 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Sepsis Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- children with sepsis, SIRS: Data will be collected and analyzed from childrens with SIRS or septic state who will be admitted to the Department of Anesthesia and Intensive Care of the University Children´s Hospital Brno, Czech Republic. Infections, sepsis, severe sepsis, septic shock and multiple organ dysfunction syndrome (MODS) will be defined according to commonly used criteria - by International pediatric sepsis consensus conference.
  Interventions: Other: therapy sepsis
- control group, healthy children: The samples children undergoing elective surgery will be used as a controls, i.e. samples from patients without signs of infection.

INTERVENTIONS:
Other: therapy sepsis — Treatment of sepsis varies depending on the site and cause of the initial infection, the organs affected and the extent of any damage
  Groups: children with sepsis, SIRS

SUMMARY:
Presepsin (formerly CD14), is a glycoprotein receptor occurring at the surface of monocytes/macrophages. CD14 binds to lipopolysaccharide (LPS) complexes and LPS binding protein (LPB), which triggers the activation of toll-like receptor 4 (TLR4), resulting in the production of numerous pro-inflammatory cytokines. Following Presepsin activation by bacterial products, the CD14 complex is released in the circulation as its soluble form (sCD14), which in turn is cleaved by a plasma protease to generate a sCD14 fragment called sCD14-subtype (sCD14- ST). Plasma levels of sCD14 can be measured using an automated chemo-luminescent assay (PATHFAST).

DETAILED DESCRIPTION:
Severe sepsis and septic shock represent major challenges of modern intensive care medicine, and still recently published international guidelines demand ongoing research about the pathophysiology, diagnostics and treatment. Currently, the diagnosis of sepsis is based on the presence of systemic inflammatory response syndrome (SIRS) criteria in the presence of a known infection. However, non-infectious SIRS associated with acute tissue injury and innate immune activation can induce clinical syndromes analogous to sepsis, including multiple trauma, pancreatitis, burns, and autoimmune diseases.

Within the field of infectious diseases, a biomarker may be used for identifying a high risk group or predisposing condition, as an aid to identification of the disease, or to direct therapy and stratify patients according to their specific risk factors, and/or as an aid to therapeutic management in order to avoid relapse of infection. Within the recent years, dozens of potential biomarkers of infection have been described. The diagnostic performance of biomarkers is usually measured in terms of sensitivity, specificity, and by likelihood ratios and area under the ROC (Receiver Operating Characteristics) curves.

Recently, several researches devolved their interest in discovering pathways involved in the innate immunity. Mediators involved in the recognition and elimination of bacterial endotoxins have been identified as new candidate biomarkers of sepsis, namely lipopolysaccharide binding protein (LBP) and soluble fractions of the membrane cluster of differentiation 14 (mCD14). Membrane CD14 is a multifunctional glycosylphosphatidylinositol-anchored membrane protein (cell surface glycoprotein), constitutively expressed by various cells, including monocytes, macrophages, neutrophils, etc. CD14 is a pattern recognition receptor for bacterial molecules, namely lipopolysaccharides (LPS) from Gram-negative bacteria and peptidoglycans together with lipoteichoic acid from Gram-positive bacteria. CD14 is crucial in activating the toll-like receptor 4 (TLR4)-specific proinflammatory signaling cascade and ultimately, initiating the inflammatory reaction against invading microorganisms. In the course of inflammatory reaction, plasma protease activity generates soluble CD14 fragments (sCD14), presepsin.

ELIGIBILITY:
Sepsis/SIRS Patients

Inclusion Criteria:

* children aged 1 - 216 months
* clinical data to enable classification into sepsis or SIRS
* written informed consent by the legally authorized representative

Exclusion Criteria:

* no informed consent

Control

Inclusion Criteria:

* children aged 1 - 216 months
* does not meet clinical criteria for sepsis or SIRS
* written informed consent by the legally authorized representative

Exclusion Criteria:

* no informed consent

Ages: 1 Month to 216 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Childrens with SIRS or septic state who will be admitted to the Department of Anesthesia and Intensive Care of the University Children´s Hospital Brno, Czech Republic. Infections, sepsis, severe sepsis, septic shock and multiple organ dysfunction syndrome (MODS) will be defined according to commonly used criteria - by International pediatric sepsis consensus conference. The samples from children undergoing elective surgery will be used as a controls, i.e. samples from patients without signs of infection.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of presepsin | up to 36 months
  Assessed the presepsin diagnostic accuracy of presepsin in diagnosing children sepsis and in discriminating systemic inflammatory response syndrome (SIRS) from sepsis. Diagnostic accuracies presented as area under the curve (AUC) for sCD14-ST.

SECONDARY OUTCOMES:
Prognostic value of presepsin | up to 36 months
  Preliminary reports suggest that levels of presepsin are significantly higher in septic patients than in healthy individuals. The aim of this study is to investigate the diagnostic and prognostic value of presepsin compared to other inflammatory markers in children with SIRS and suspected sepsis or septic shock. Receiver operating characteristic (ROC) curve analysis will performed for presepsin and compared to ROC curve analysis of current available infection biomarkers.

OTHER OUTCOMES:
Mortality | up to 36 months
  Sepsis mortality in children remains high despite advances in diagnosis and treatment. Early identification and risk stratification is a key point in the triage of patients with sepsis. The aim of the study is identifying and testing of presepsin with improved sensitivity and specifity for the presence of sepsis, and prediction of morbidity and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Žurek, M.D., Ph.D., Principal Investigator — Department of Anesthesia and Intensive Care, University Children´s Hospital
Locations (1):
- Faculty Hospital Brno, Brno, Czechia